CLINICAL TRIAL: NCT06373757
Title: Chitosan Nano-hydroxyapatite Hydrogel in Non-Surgical Treatment of Intrabony Defect (Randomized Clinical Trial)
Brief Title: Chitosan Nano-hydroxyapatite Hydrogel in Non-Surgical Treatment of Intrabony Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amany Ahmed Mohamed Alaraby, Lecturer of Oral Medicine, Diagnosis and Periodontology Department, Faculty of Dentistry, October 6 University, 6 October city, Egypt, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECO6U/5-2023
Record Dates: First submitted 2024-04-09; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Chitosan; Nano-hydroxyapatite Hydrogel; Intrabony Defect

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (nano-HAP/Chitosan hydrogel): (Experimental): The periodontal pockets more than or equal 3-5mm were isolated. Chitosan and nano-HAP hydrogel were prepared in the same steps that were mentioned in the methodology and then the prepared gel was applied to the test site of patients with the deepest probing pocket measurement once per week for 3 weeks. Periodontal dressing (Coe-pack) was to secure the hydrogel in place.
  Interventions: Other: Nano-HAP/Chitosan hydrogel
- Group II (No Intervention): Patients were treated with supra and sub-gingival debridement only.

INTERVENTIONS:
Other: Nano-HAP/Chitosan hydrogel — The periodontal pockets more than or equal 3-5mm were isolated. Chitosan and nano-HAP hydrogel were prepared in the same steps that were mentioned in the methodology and then the prepared gel was applied to the test site of patients with the deepest probing pocket measurement once per week for 3 weeks. Periodontal dressing (Coe-pack) was to secure the hydrogel in place.
  Arms: Group I (nano-HAP/Chitosan hydrogel):

SUMMARY:
The aim of this study was to evaluate the clinical effect of Chitosan with nano-hydroxyapatite hydrogel in the treatment of periodontal intrabony defects.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammation of the periodontium that extends beyond the gingiva and involves the destruction of the connective tissue attachment of the teeth.

Treatment modalities of periodontitis includes local drug delivery such as chitosan which is a derivative of the exoskeleton of many arthropods including prawns, lobsters and crabs.

Chitosan has been used in guided bone regeneration, hemostasis of surgical wounds, and coating of dental implants, in reconstruction of temporomandibular joint disc and guided periodontal tissue regeneration. Moreover, chitosan has been used for preventing demineralization.

HA also called hydroxylapatite, is a naturally occurring mineral form of calcium apatite with the formula Ca5(PO4)3(OH). The OH- ion can be replaced by fluoride, and carbonate, producing fluorapatite or chlorapatite. It crystallizes in the hexagonal crystal system.

ELIGIBILITY:
Inclusion Criteria:

* Age from 25 to 55 years.
* Both sexes.
* Patients with stage II to III periodontitis with probing pocket depths ≥ 5 mm and radiographic evidence showing infrabony defect.

Exclusion Criteria:

* Patients received periodontal or antibiotic therapy within the previous 6 months preceding the study.
* Smokers.
* Pregnant and lactating females.
* Patients on medications known to affect bone turnover or with known side effects to chitosan, nano-hydroxyapatite, and collagen membrane.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Gingival index | 6 months after treatment
  Gingival index (GI) used for the assessment of prevalence and severity of gingivitis. A score from 0 to 3 is given to each area of the tooth.0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation from, and 2.1-3.0 signifies severe inflammation.
  It was evaluated for every patient included in the study, 3 and at 6 months after treatment.

SECONDARY OUTCOMES:
Plaque index | 6 months after treatment
  Plaque index (PI) was used to assess oral hygiene where 0 = no plaque. 1 = separate flecks of plaque at the cervical margin of the tooth. 2 = a thin continuous band of plaque (up to 1 mm) at the cervical margin of the tooth.
  It was evaluated for every patient included in the study, 3 and at 6 months after treatment.
Clinical attachment level | 6 months after treatment
  Clinical attachment level (CAL) was evaluated for every patient included in the study, 3 and at 6 months after treatment.
Periodontal probing depth | 6 months after treatment
  Periodontal probing depth (PD) (referred to as pocket depth if periodontal disease is present) is the distance from the gingival margin to the apical portion of the gingival sulcus. Probing depths in healthy gingival sulci normally range from 1 to 3 mm.
  It was evaluated for every patient included in the study, 3 and at 6 months after treatment.
Acrylic stent for pocket assessment | 6 months after treatment
  Acrylic stent for pocket assessment was evaluated for every patient included in the study, 3 and at 6 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.